CLINICAL TRIAL: NCT03877913
Title: Daily ECG Transmission Versus Serial 7-day Holter ECG for Assessment of Efficacy of Ablation for Atrial Fibrillation - the AGNES-ECG Study
Brief Title: Daily ECG Versus 7-day Holter ECG After Atrial Fibrillation Ablation
Acronym: AGNES-ECG
Status: Completed | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Prof. Piotr Kulakowski, professor, Centre of Postgraduate Medical Education
Other Study IDs: 86/PB/2018
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; electrocardiographic monitoring
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction:

The optimal method for the assessment of efficacy of ablation for atrial fibrillation (AF) has not yet been established. The symptom-based evaluation is not accurate because many AF episodes are asymptomatic. It has been well documented that the more frequent and/or longer ECG recording the more the AF recurrences are detected. However, such devices for long-term ECG monitoring as implantable loop recorders are expensive whereas external ECG monitoring is not well tolerated over a period longer than one month. The most frequently used approach is periodic 1-7 day Holter ECG monitoring, usually performed 3, 6 and 12 months after the procedure and additional standard ECG recordings when symptoms occur. Using this method, asymptomatic AF episodes occurring between Holter ECG recordings are missed.

Recently, several types of external ECG recorders have been introduced, enabling good quality frequent ECG recordings and transmission via mobile phones. Only a few studies documented the usefulness of this method in detecting silent AF in a high-risk population, however, the value of short but frequent ECG recordings after AF ablation has not yet been established. In these studies, short ECG recordings performer once or twice daily detected the highest number of AF episodes.

In summary, data on the optimal type of ECG monitoring after AF ablation are scarce. It seems that frequent, short ECG recordings have more diagnostic yield than 24-hour ECG monitoring, even when performed monthly, or standard care with recording ECG only when symptoms suggesting AF occur. However, the optimal mode of monitoring is not known. Such questions as whether once-a-day ECG transmission is enough and whether longer i.e. 7-day Holter ECG may be as valuable as daily ECG transmissions, remain unanswered.

Aim: to compare daily ECG transmissions with repeated 7-day Holter ECG in detecting AF episodes following AF ablation.

Hypothesis: daily ECG recordings have significantly higher yield in AF detection than repeated 7-day Holter ECG.

Methods:

The study group will consists of 50 consecutive patients undergoing AF ablation in the investigator's center. Only patient capable of maintain ISTEL recorder and transmitting ECG will be enrolled in the study (1-2 day after catheter ablation for AF). The follow-up will last 12 months. The AF detection will be performed using two recording methods in each patient. The number of 50 patients has been chosen based on the assumption that Holter ECG will detect AF recurrence in 15% of patients and daily transmission will detect AF recurrence in 38% patients (alfa error = 0.05 and beta error = 0.2).

Daily ECG recordings and transmissions will be performed using the HR-2000 recorder (ISTEL, Poland). This device enables recording of 30 seconds of 6-channel ECG (I, II, III, aVR, aVL, aVF) from 4 metal electrodes build in the recorder. In order to record ECG, the device is activated by a patient and attached to the thorax, at the area of sternum. The duration of recording may vary from 30 seconds to 3 minutes, however, only 30-second recordings will be used in the present study. After recording, ECG will be transmitted using Bluetooth to patient's smartphone and then transmitted to the central station where they will be stored and analyzed. Analysis will be performed on a daily basis by an experienced ECG technician, not directly involved in patient's recruitment and treatment. The results of all recordings will be available for study team after 3, 6 and 12 months after ablation, at the time when concurrent Holter ECG recordings will be analyzed. Only in case of serious, life-threatening arrhythmias (non-sustained or sustained ventricular tachycardia, or pauses > 6 seconds) the study team will be informed immediately by a technician about the results of 30-second ECG recording in order to undertake proper action. Specifically, asymptomatic episodes of AF will not be unblinded to the study team in order not to interfere with medication and to allow continuing follow-up till next Holter ECG monitoring.

The second method of ECG recording will be 7-day Holter ECG (DMS 300-4A recorders, DM Software, NV, USA) performed 3, 6 and 12 months after ablation.

The patients will be allowed to record additional ECG when symptoms suggesting AF occur. This may be performed by ISTEL recorder or standard 12-lead ECG if available.

At each time-point (3, 6 and 12 months) the study team will analyze all recorded ECGs and 7-day Holter ECG, and make appropriate therapeutic decisions.

Anticipated results:

* Daily ECG recordings will detect first AF episode faster than standard Holter monitoring.
* ISTEL recorder will identify more patients with AF recurrence than standard Holter monitoring
* ISTEL recorder will identify more patients with asymptomatic AF recurrence than standard Holter monitoring

Definitions:

AF episode - episode lasting ≥30 seconds Study period: August 2018 - August 2020

DETAILED DESCRIPTION:
Daily ECG transmission versus serial 7-day Holter ECG for assessment of efficacy of ablation for atrial fibrillation - the AGNES-ECG study

Introduction. The optimal method for the assessment of efficacy of ablation for atrial fibrillation (AF) has not yet been established. The symptom-based evaluation is not accurate because many AF episodes are asymptomatic. It has been well documented that the more frequent and/or longer ECG recording the more the AF recurrences are detected. However, such devices for long-term ECG monitoring as implantable loop recorders are expensive whereas external ECG monitoring is not well tolerated over a period longer than one month. The most frequently used approach is periodic 1-7 day Holter ECG monitoring, usually performed 3, 6 and 12 months after the procedure and additional standard ECG recordings when symptoms occur [1]. Using this method, asymptomatic AF episodes occurring between Holter ECG recordings are missed.

Recently, several types of external ECG recorders have been introduced, enabling good quality frequent ECG recordings and transmission via mobile phones. Only a few studies documented the usefulness of this method in detecting silent AF in a high-risk population [2], however, the value of short but frequent ECG recordings after AF ablation has not yet been established. Kimura et al. [3] tested three methods for AF detection after ablation in 30 patients. The follow-up lasted 6 months and each patient underwent three types of ECG recordings (1) repeated 10-second standard ECG recordings, obtained during outpatient visits, (2) 24-hour Holter ECG performed every month and (3) short 30-second ECG recordings performed twice daily and when symptoms occur, transmitted by telemetry. As expected, the latter method enabled detection of the highest number of AF episodes, however, the number of recordings declined steadily throughout the period of the study, suggesting some technical difficulties with performing recordings and decreased patient compliance.

Similar study was conducted by Senatore et al. [4] who compared diagnostic yield of twice daily ECG tele-transmission versus repeated 24 hour ECG recordings in 72 patients after AF ablation. Using daily ECG transmissions, significantly more patients had AF episodes detected (27.8% vs 13.9%, p = 0,001). In another study [5] twice daily ECG transmissions using smartphone and AliveCor system were compared with standard medical care in patients with a history of AF undergoing ablation or cardioversion. Also in this study frequent ECG transmissions using smartphone occurred more effective in detecting AF recurrences than standard care (61% vs 30%; P = 0,04).

In summary, data on the optimal type of ECG monitoring after AF ablation are scarce. It seems that frequent, short ECG recordings have more diagnostic yield than 24-hour ECG monitoring, even when performed monthly, or standard care with recording ECG only when symptoms suggesting AF occur. However, the optimal mode of monitoring is not known. Such questions as whether once-a-day ECG transmission is enough and whether longer i.e. 7-day Holter ECG may be as valuable as daily ECG transmissions, remain unanswered.

Aim: to compare daily ECG transmissions with repeated 7-day Holter ECG in detecting AF episodes following AF ablation.

Hypothesis: daily ECG recordings have significantly higher yield in AF detection than repeated 7-day Holter ECG.

Methods:

Patients:

The study group will consists of 50 consecutive patients undergoing AF ablation in the investigator's center. The follow-up will last 12 months. The AF detection will be performed using two recording methods in each patient. The number of 50 patients has been chosen based on the assumption that Holter ECG will detect AF recurrence in 15% of patients and daily transmission will detect AF recurrence in 38% patients (alfa error = 0.05 and beta error = 0.2)

Daily ECG recordings and transmissions will be performed using the HR-2000 recorder (ISTEL, Poland). This device enables recording of 30 seconds of 6-channel ECG (I, II, III, aVR, aVL, aVF) from 4 metal electrodes build in the recorder. In order to record ECG, the device is activated by a patient and attached to the thorax, at the area of sternum. The duration of recording may vary from 30 seconds to 3 minutes, however, only 30-second recordings will be used in the present study. After recording, ECG will be transmitted using Bluetooth to patient's smartphone and then transmitted to the central station where they will be stored and analyzed. Analysis will be performed on a daily basis by an experienced ECG technician, not directly involved in patient's recruitment and treatment. The results of all recordings will be available for study team after 3, 6 and 12 months after ablation, at the time when concurrent Holter ECG recordings will be analyzed. Only in case of serious, life-threatening arrhythmias (non-sustained or sustained ventricular tachycardia, or pauses > 6 seconds) the study team will be informed immediately by a technician about the results of 30-second ECG recording in order to undertake proper action. Specifically, asymptomatic episodes of AF will not be unblinded to the study team in order not to interfere with medication and to allow continuing follow-up till next Holter ECG monitoring.

The second method of ECG recording will be 7-day Holter ECG (DMS 300-4A recorders, DM Software, NV, USA) performed 3, 6 and 12 months after ablation.

The patients will be allowed to record additional ECG when symptoms suggesting AF occur. This may be performed by ISTEL recorder or standard 12-lead ECG if available.

At each time-point (3, 6 and 12 months) the study team will analyze all recorded ECGs and 7-day Holter ECG, and make appropriate therapeutic decisions.

Inclusion criteria

1. AF ablation 1-3 days prior to inclusion
2. Access to smartphone and ability to maintain ISTEL recorder and transmitting ECG.

Exclusion criteria.

1. Pacemaker implanted.
2. Known presence of other than AF cardiac arrhythmias requiring frequent ECG monitoring (ventricular arrhythmia, second or third-degree atrioventricular block)
3. Lack of smartphone or inability to manage ISTEL recorder.

1. Primary end-point: Time to detection of first AF episode after ablation 2. Secondary end-point: Number of patients with AF recurrence after ablation Number of patients with asymptomatic AF recurrence after ablation

Definitions AF episode - episode lasting ≥30 seconds Study period: August 2018 - August 2020

ELIGIBILITY:
Inclusion Criteria:

1. AF ablation 1-3 days prior to inclusion
2. Access to smartphone and ability to maintain ISTEL recorder and transmitting ECG.

Exclusion Criteria:

1. Pacemaker implanted.
2. Known presence of other than AF cardiac arrhythmias requiring frequent ECG monitoring (ventricular arrhythmia, second or third-degree atrioventricular block)
3. Lack of smartphone or inability to manage ISTEL recorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing standard abaltion for AF
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Time to first AF episode recurrence | one year
  Time in days to first AF episode recurrence documented by either of studied methods

SECONDARY OUTCOMES:
Number of patients with AF episodes | one year
  Number of patients with AF episode recurrence documented by either of studied methods
Number of patients with asymptomatic AF episodes | one year
  Number of patients with asymptomatic AF episode recurrence documented by either of studied methods

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kulakowski, MD, Principal Investigator — Centre of Postgraduate Medical Education; Agnieszka Sikorska, MD, Principal Investigator — Centre of Postgraduate Medical Education
Locations (1):
- Centre of Postgraduate Medical Education, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed, raw data will be available to other investigators
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From August 2020
Access Criteria: contact by mail

REFERENCES:
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Cosedis Nielsen J, Curtis AB, Davies DW, Day JD, d'Avila A, Natasja de Groot NMS, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T; Document Reviewers:. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Europace. 2018 Jan 1;20(1):e1-e160. doi: 10.1093/europace/eux274. No abstract available. PMID 29016840
- [Result] Halcox JPJ, Wareham K, Cardew A, Gilmore M, Barry JP, Phillips C, Gravenor MB. Assessment of Remote Heart Rhythm Sampling Using the AliveCor Heart Monitor to Screen for Atrial Fibrillation: The REHEARSE-AF Study. Circulation. 2017 Nov 7;136(19):1784-1794. doi: 10.1161/CIRCULATIONAHA.117.030583. Epub 2017 Aug 28. PMID 28851729
- [Result] Kimura T, Aizawa Y, Kurata N, Nakajima K, Kashimura S, Kunitomi A, Nishiyama T, Katsumata Y, Nishiyama N, Fukumoto K, Tanimoto Y, Fukuda K, Takatsuki S. Assessment of atrial fibrillation ablation outcomes with clinic ECG, monthly 24-h Holter ECG, and twice-daily telemonitoring ECG. Heart Vessels. 2017 Mar;32(3):317-325. doi: 10.1007/s00380-016-0866-2. Epub 2016 Jul 6. PMID 27385021
- [Result] Senatore G, Stabile G, Bertaglia E, Donnici G, De Simone A, Zoppo F, Turco P, Pascotto P, Fazzari M. Role of transtelephonic electrocardiographic monitoring in detecting short-term arrhythmia recurrences after radiofrequency ablation in patients with atrial fibrillation. J Am Coll Cardiol. 2005 Mar 15;45(6):873-6. doi: 10.1016/j.jacc.2004.11.050. PMID 15766823
- [Result] T Hickey K, B Biviano A, Garan H, Sciacca RR, Riga T, Warren K, Frulla AP, Hauser NR, Wang DY, Whang W. Evaluating the Utility of mHealth ECG Heart Monitoring for the Detection and Management of Atrial Fibrillation in Clinical Practice. J Atr Fibrillation. 2017 Feb 28;9(5):1546. doi: 10.4022/jafib.1546. eCollection 2017 Feb-Mar. PMID 29250277
- [Derived] Sikorska A, Baran J, Piotrowski R, Krynski T, Szymot J, Soszynska M, Kulakowski P. Daily ECG transmission versus serial 6-day Holter ECG for the assessment of efficacy of ablation for atrial fibrillation - the AGNES-ECG study. J Interv Card Electrophysiol. 2022 Nov;65(2):373-380. doi: 10.1007/s10840-022-01166-4. Epub 2022 Mar 3. PMID 35244820